CLINICAL TRIAL: NCT02418767
Title: A Randomized, Double-blind, Vehicle-controlled, Parallel Group, Single Dose Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Three Doses of Long Acting HGH Product (MOD-4023) in Healthy Caucasian and Japanese Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of Long Acting Human Growth Hormone (hGH) Product (MOD-4023) in Healthy Caucasian and Japanese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CP-4-007
Record Dates: First submitted 2015-01-08; First posted 2015-04-16 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — MOD-4023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low dose (Experimental): 7 Japanese and 7 Caucasian subjects (randomized 6:1) administered a single dose of MOD-4023/Placebo
  Interventions: Drug: MOD-4023; Drug: Placebo
- Mid dose (Experimental): 7 Japanese and 7 Caucasian subjects (randomized 6:1) administered a single dose of MOD-4023/Placebo
  Interventions: Drug: MOD-4023; Drug: Placebo
- High dose (Experimental): 7 Japanese and 7 Caucasian subjects (randomized 6:1) administered a single dose of MOD-4023/Placebo
  Interventions: Drug: MOD-4023; Drug: Placebo

INTERVENTIONS:
Drug: MOD-4023
Drug: Placebo

SUMMARY:
The study is a Phase 1, randomized, double-blind, vehicle-controlled, single-dose, three dose levels study in healthy Caucasian and Japanese male volunteers.

Following a 4-week screening period, eligible male subjects will be stratified by ethnic group and will be randomized to one of six groups. On dosing day, designated as Day 1, each subject will receive single SC injection of study medication according to group allocation and will be followed up for a month for safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, 18 to 45 years of age (inclusive).
2. Body Mass Index (BMI) 18 to 30 kg/m2 (inclusive) and weighing at least 55 kg.
3. Subjects in generally good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
4. Blood pressure and heart rate within normal limits.
5. Electrocardiogram (ECG) with no clinically significant abnormalities recorded at screening visit (up to 28 days before dosing) and on dosing day (before drug administration).
6. Negative HIV, hepatitis B and hepatitis C serology tests at screening
7. No clinically significant abnormalities in complete blood count (CBC), international normalized ratio (INR), chemistry lab tests (liver and renal function) and urinalysis at screening.
8. No history of alcohol or drug abuse within 1 year of screening. Negative urine drugs-of-abuse (DOA) in screening and on admission. Negative breath alcohol on admission.
9. Subjects must agree to use medically accepted form of contraception from dosing day to 12 weeks after drug administration.
10. Subjects must be able to understand the requirements of the study and must be willing to comply with the requirements of the study and to provide their written informed consent to participate in the study.

Exclusion Criteria:

1. History of significant neurological (including history of seizures or EEG abnormalities), renal, cardiovascular (including known structural cardiac abnormalities or hypertension), respiratory (asthma), endocrinological, gastrointestinal, hematopoietic disease, neoplasm, psychological (marked anxiety, tension or agitation) or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medication.
2. Known allergy to growth hormone or any constituents or ingredients or components in the vehicle.
3. Adherence (for whatever reason) to an abnormal diet (including any dietary restrictions, e.g. low fat, lactose-free, low sodium, high protein, gluten-free, organic, etc.) during the 4 weeks prior to the study, or subjects with recent significant change in body weight.
4. Use of any prescription or over-the-counter (OTC) medications, including vitamins and herbal or dietary supplements within 14 days prior to dosing. Brief use of OTC medications for symptomatic relief of pain until 24 hours prior to and 48 hours after the study drug administration may be allowed per the discretion of the medical monitor.
5. Subjects who have received any vaccines within 4 weeks prior to study drug administration.
6. Subjects who donated blood or received blood or plasma derivatives in the one month preceding signing of consent form.
7. Systemic corticosteroids other than in replacement doses within the 3 months before study entry (temporary adjustment of glucocorticoids, as appropriate, is acceptable)
8. Anabolic steroids other than gonadal steroid replacement therapy within 2 months before study entry
9. Participation in another clinical trial with drugs within one month of signing of consent form (calculated from the previous study's last dosing date).
10. Subjects with an inability to communicate well with the investigators and clinic staff [i.e., language problem (except Japanese speakers), poor mental development or impaired cerebral function].
11. Subjects with any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator. Use of investigational products (within 30 days of screening visit).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Composite safety and tolerability parameters as measured by adverse events, electrocardiograms (ECG), laboratory results, vital signs and injection site reactions | 30 days
  To assess the safety, tolerability and immunogenicity of MOD-4023 in healthy Caucasian and Japanese subjects after single subcutaneous (SC) dose.
Pharmacokinetics (PK) profile of MOD-4023 in healthy Caucasian and Japanese subjects after single SC dose | 7 days
  MOD-4023 serum levels (T1/2, Area-Under-the-Curve, Cmax, Tmax)

SECONDARY OUTCOMES:
Pharmacodynamic (PD) profile (IGF-1 and IGFBP-3 levels) to MOD-4023 in healthy Caucasian and Japanese subjects after single SC dose | 14 days
  IGF-1 and IGFBP-3 serum levels (T1/2, AUC, Cmax, Tmax)

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, Cypress, California, United States